CLINICAL TRIAL: NCT07398079
Title: Pilot Observational Study of an Integrative Cure Stay Program
Acronym: Via Shalva
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-01722;bb25Heinz-Schwarz7
Record Dates: First submitted 2026-01-12; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Gynecologic Cancer
Keywords: Complementary Therapies; Integrative Medicine; Feasibility Studies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Integrative Cure Stay Group: Participants attend a 7-day integrative oncology retreat including individualized consultations, complementary therapies, and group-based mind-body interventions.
  Interventions: Behavioral: Integrative Cure Stay
- Matched Control Group: Participants receive usual oncology follow-up without attending the retreat.
  Interventions: Other: Matched Control Group

INTERVENTIONS:
Behavioral: Integrative Cure Stay — Participants attend a 7-day integrative oncology retreat including individualized consultations, complementary therapies, and group-based mind-body interventions
  Groups: Integrative Cure Stay Group
Other: Matched Control Group — Participants receive usual oncology follow-up without attending the retreat
  Groups: Matched Control Group

SUMMARY:
This pilot observational study evaluates the feasibility and acceptability of conducting a prospective study alongside the individualized integrative oncology cure stay program "Via Shalva" for breast and gynecological cancer survivors. The study further explores preliminary changes in patient-reported outcomes, physiological measures, and biological markers before and after the retreat and compared with a matched control group.

DETAILED DESCRIPTION:
Breast and gynecological cancer survivors frequently experience long-term physical and psychological symptoms after completing primary treatment, including fatigue, anxiety, stress, sleep disturbances, and reduced quality of life. Integrative oncology approaches-such as acupuncture, yoga, mindfulness, psycho-oncological support, and individualized lifestyle counselling-may help alleviate these symptoms, but evidence from structured, prospective research remains limited. "Via Shalva," a 7-day integrative oncology retreat, was developed to address these unmet supportive care needs.

This prospective, exploratory, single-center observational matched cohort study aims to evaluate the feasibility of conducting a clinical study alongside the retreat, including recruitment, retention, adherence, and completeness of data collection. Participants attending the cure stay are compared with a matched control group not participating in the retreat. Study procedures include systematic assessment of patient-reported outcomes, wearable-based physiological data, and biological samples. Measurements are performed longitudinally across six time points over six months.

Secondary exploratory aims include describing potential changes in symptoms, wellbeing, and stress-related biomarkers following the retreat, as well as differences between retreat participants and controls. Findings will inform the design of future randomized controlled trials evaluating integrative oncology interventions and contribute to improving supportive cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Breast and gynecological cancer (including but not limited to ovarian, endometrial, cervical, vulvar and vaginal cancer) survivors, including recurrent disease
* Completed primary treatment (operation +/- radiation +/- chemotherapy)
* Age ≥ 18 years
* Ongoing or planned maintenance treatment scheduled for > 3 months during study period is allowed (e.g. antihormonal therapy, Anti-Her2-antibodies, CDK4/6-inhibitors, Anti-VEGF-inhibitor, PARP-inhibitor, immune-checkpoint inhibitors etc.)
* Signed informed consent for participation of the trials
* Presence of a stoma is allowed
* Prior cancer is allowed
* Prior treatment - including chemotherapy - for a prior malignant tumor (including breast or gynecological cancer) is allowed
* Concomitant participation in an experimental therapeutic drug trial is allowed
* Use of other complementary methods (including mistletoe) is allowed
* Pregnancy is allowed.

Exclusion Criteria:

* Language or cognitive deficits (including impaired consciousness) that are incompatible with the participation in the study
* Severe physical or psychiatric comorbidity that prevents a patient from participating in the study
* Patients incapable of giving consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast and gynecological cancer survivors who have completed primary treatment (surgery ± chemotherapy ± radiotherapy) and continue to experience long-term physical or psychological symptoms.
  A matched control group consists of similar patients not attending the integrative cure stay program.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Study Conduct (Composite Outcome) | Baseline to 6 months
  Feasibility of study conduct assessed as a composite outcome based on predefined feasibility criteria, including recruitment rate, retention rate, adherence to study procedures, completeness of data collection, and logistical/operational feasibility. Overall feasibility will be determined by whether predefined thresholds for these criteria are met.

SECONDARY OUTCOMES:
Quality of Life (EQ-5D-5L) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in health-related quality of life measured using the EQ-5D-5L questionnaire. EQ-5D-5L scoring involves combining responses from 5 dimensions (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression) into a 5-digit profile with values ranging from 11111 (best possible health state) to 55555 (worst possible health state). A separate EQ Visual Analog Scale (VAS) provides a subjective "health today" score (0-100).
Quality of Life (VAS) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  The EQ Visual Analog Scale (VAS) provides a subjective "health today" score (0-100).
Psychological Distress (Distress Thermometer) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in psychological distress assessed using the Distress Thermometer, a valid and reliable measure developed by the National Comprehensive Cancer Network for screening psychological distress in cancer patients. The German version was adapted by Mehnert et al. A score of 5 or higher at the visual analogue scale. The score ranges from 0-10 while 10 indicates a higher stress level.
Perceived Stress (PSS-10) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in perceived stress levels measured with the 10-item Perceived Stress Scale. PSS-10 measures the degree to which life has been perceived as unpredictable, uncontrollable und overloading over the last month. The responses are rated on a 5-point rating scale with a total score ranging from 0-40 while a higher total score indicating greater stress.
Anxiety and Depression (HADS) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in anxiety and depression symptoms measured by the Hospital Anxiety and Depression Scale.
  The scale consists of 14 questions, with each question being assigned a value from 0 to 3. The total score can range from 0 to 21. Scores of 8-10 are considered borderline, 11-15 moderate, and 16 or higher severe anxiety or depression.
Resilience (CD-RISC-10) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in psychological resilience measured using the CD-RISC-10 questionnaire. It is the shortened version of a 25-items questionnaire which evaluates the patient's ability to bounce back when diagnosed with a disease. The responses are rated on a 5-point rating scale with the total score ranged from 0-40 while a higher total score indicating greater resilience.
Therapy Adherence | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in adherence to ongoing maintenance therapies assessed via routine visit documentation and follow-up questionnaires.
Physiological Measures: HRV | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in heart rate variability using a wearable device.
Physiological Measures (Pulse) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in pulse measured using a wearable device.
Physiological Measures (physical activity) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change of daily physical activity is evaluated by the number of steps using a wearable device.
Salivary Cortisol | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in diurnal cortisol levels (awakening, +30 min, +1 h, +6 h, +14 h) measured by LC-MS/MS.
Salivary Alpha-Amylase (sAA) | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in salivary alpha-amylase activity as a biomarker of sympathetic activation.
Serum BDNF | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Change in serum brain-derived neurotrophic factor levels measured via ELISA.
Microbiome Composition | Baseline, pre-retreat, last day of retreat, 2 weeks, 1 month, 3 months, 6 months.
  Exploratory changes in gut, oral, and urinary microbiome diversity and composition assessed by 16S rRNA sequencing.
Subjective Evaluation of the Cure Stay | Daily from day 3 to day 7 of the cure stay
  Participants' satisfaction and perceived benefit of the integrative cure stay is assessed by the questionnaire "personal evaluation of the cure stay". Scores ranges from 0-24 while higher scores indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Viola Heinzelmann-Schwarz, Prof. MD, Study Chair — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No